CLINICAL TRIAL: NCT05056519
Title: A Random, Double -Blind, Placebo Control Phase Ⅰ Trail to Evaluate the Safety and Immunogenicity of Live Attenuated Influenza Vaccine in 3-59y Healthy People
Brief Title: The Safety and Immunogenicity Evaluation of Live Attenuated Influenza Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Collaborators: He Bei province Center for Disease control and prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: F20210719
Record Dates: First submitted 2021-08-31; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Influenza Prevention
Keywords: Safety; Immunogenicity; Live Attenuated Influenza Vaccine
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Totally 160 in 3-59 years old healthy people will be divided into two age group, which contain 80 people in 18-59 years old and 80 people in 3-17 years old. In each age group, subjects will be randomly divided into vaccine group and placebo group in a ratio of 3:1.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The design of this trail is based on random, two-blind, placebo control. The subjects and investigators will not know the masking status, unless the specific subjects who required treatment for serious adverse events .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Healthy people in experimental group will receive a dose of Live Attenuated Influenza Vaccine
  Interventions: Biological: Live Attenuated Influenza Vaccine
- Placebo group (Placebo Comparator): Healthy people in placebo group will receive a dose of placebo
  Interventions: Biological: Live Attenuated Influenza Vaccine placebo

INTERVENTIONS:
Biological: Live Attenuated Influenza Vaccine — Live Attenuated Influenza Vaccine placebo, containing H1, H3 and B type influenza Live Attenuated virus.
  Arms: Experimental group
Biological: Live Attenuated Influenza Vaccine placebo — Live Attenuated Influenza Vaccine placebo, not containing H1, H3 and B type influenza Live Attenuated virus.
  Arms: Placebo group

SUMMARY:
Live Attenuated freeze-dried Influenza Vaccine has been licensed for use in 2020 (Approval No.S20200002), the sponsor of this research submitted an new application for non freeze-dried Live Attenuated Influenza Vaccine in 2021. The main objective of phase Ⅰ trail is to evaluate the safety of LAVI(non freeze-dried). The secondary objective is to evaluate the immunogenicity of LAVI(non freeze-dried).

DETAILED DESCRIPTION:
Totally 160 health people aged 3-59 years old will be divided into two age group, containing 80 in 18-59 years old and 80 in 3-19 years old. All subjects will receive vaccination either LAVI or placebo in a ratio of 3:1.

All subjects will be collected any adverse events within 30 days and any serious adverse events within 6 months for safety evaluation.

All subjects will be collected blood sample and nasopharyngeal swab for immunogenicity evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged in 3-59 years old.
* Had not received vaccination of Influenza vaccine in the past half of years.
* Had not infected with Influenza virus.
* This trail has been agreed by volunteers or his/her legal guardian.
* Volunteers or his/her legal guardian will fellow this trail protocol.

Exclusion Criteria:

* People from 18-59 age group with abnormal laboratory index. (slight abnormality is except if judged with no clinical significance by doctors.)
* People with fever before vaccination, temperature higher than 37.0 ℃
* Females in suckling period, pregnancy (pregnancy test positive) or prepared to be pregnant
* People given whole blood, plasma or immunoglobulin therapy within 3 months before vaccination
* According to judgement of researchers, the subjects have any other factors that are not appropriate for this clinical trials.
* Acute infectious disease or acute attack of chronic disease before inoculation
* People get any vaccine within 14 days before the trial.
* People in immune deficiency or diagnosed with congenital or acquired immunodeficiency, people with immunosuppressive therapy in the past six months.
* People with epilepsy or a history of mental illness

Ages: 3 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as assessed by SAS v9.4 | Within 31 days after vaccination
  The incidence rate of adverse events in all subjects
Number of participants with laboratory examination abnormity as assessed by SAS v9.4Clinical laboratory examination | 3 days after vaccination
  The incidence rate of abnormal of Blood routine, blood biochemical and urine in The incidence rate of abnormality of blood routine, blood biochemical and urine routine in 18-59 years age group
Number of participants with virus Shedding as assessed by SAS v9.4 | within 16 days after vaccination
  The nasal secretions of Subjects in 18-59 years age group will be taken and be tested

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Provincial Center for Disease Control and Prevention, Shijiazhuang, Hebei, China